CLINICAL TRIAL: NCT07392151
Title: REVERsal to Normoglycemia by Treating PREDIABETES: The REVERT-PREDIABETES Trial
Brief Title: Reversal to Normoglycemia by Treating Prediabetes
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Michael Mæng (Other)
Collaborators: Aarhus University Hospital (Other); GCP-unit at Aarhus University Hospital, Aarhus, Denmark (Other); Department of Clinical Epidemiology, Aarhus University, DK-8200 Aarhus N, Denmark (Unknown); University of Aarhus (Other); Steno Diabetes Center Aarhus (SDCA), Aarhus University Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Michael Mæng, MD, PhD, Professor, FESC, Aarhus University Hospital Skejby
Organization: Aarhus University Hospital Skejby (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025-522970-35-00
Record Dates: First submitted 2026-01-23; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Prediabetes; Chronic Coronary Syndrome
Keywords: Prediabetes; Chronic coronary syndrome; Coronary artery disease; Normoglycemia; Semaglutide; Dapagliflozin; Retinopathy; Neuropathy; Nephropathy; MASLD
MeSH Terms: conditions — Prediabetic State; Coronary Artery Disease; Retinal Diseases; Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Prediabetes: Interventional therapy arm (Experimental): Intensified medical follow-up and treatment including cardioprotective glucose-lowering drugs
  Interventions: Drug: Intensified medical follow-up and glucose-lowering drugs
- Prediabetes: Conventional therapy arm (No Intervention): Current practice
- Normoglycemia (Other): Baseline comparator group
  Interventions: Other: No intervention

INTERVENTIONS:
Drug: Intensified medical follow-up and glucose-lowering drugs — Intensified medical follow-up and treatment including cardioprotective glucose-lowering drugs
  Arms: Prediabetes: Interventional therapy arm
Other: No intervention — Baseline comparator group
  Arms: Normoglycemia

SUMMARY:
Prediabetes is a precursor to diabetes, but compared with diabetes, much less is known about prediabetes. Prediabetes is defined based on a blood sample measuring long-term average glucose levels. In the Danish population, about 7% have prediabetes, and roughly one in five will develop diabetes within five years. In the US, significantly more people have this condition - about 38% of the adult population - and it is reasonable to expect a growing global prevalence over the years.

Diabetes is associated with various microvascular diseases, traditionally referred to as diabetic complications, such as diabetic retinopathy, diabetic nephropathy, and diabetic neuropathy. However, it has been shown that some of these conditions are already present in some individuals with prediabetes, even though this condition does not meet the diagnostic criteria for diabetes. Several metabolic changes are often seen in people with prediabetes, including high cholesterol, hypertension, increased inflammatory markers, and obesity. Additionally, there is a possible link between prediabetes and the occurrence of fat accumulation in the liver. These risk factors are also believed to be associated with the development of coronary atherosclerosis. In individuals with coronary atherosclerosis there is an overrepresentation of prediabetes. Therefore, the investigators would like to investigate whether this group of people might benefit from having their long-term average glucose levels reduced to normal from prediabetes using glucose-lowering medication, which is approved for use in people with diabetes and has also shown a cardioprotective effect in individuals without diabetes.

The medications that will be used for this purpose are:

Semaglutide, administered once weekly as a subcutaneous injection. The dose will be gradually increased at 4-week intervals up to a maximum of 2.4 mg. If this is insufficient, it may be considered to start Dapagliflozin (Forxiga), 10 mg tablet daily. Both treatments are approved for use in Europe but are not currently used to treat prediabetes.

A total of 108 individuals with prediabetes and coronary atherosclerosis who consent to participate in the trial will be randomly assigned (1:1) to two groups:

1. Interventional therapy arm: Participants will attend visits at Aarhus University Hospital and begin glucose-lowering treatment. Additionally, any hypertension or high cholesterol will be optimized according to current guidelines. They will be offered lifestyle counselling. Participants will have their blood pressure measured regularly and, if necessary, blood samples are drawn to optimize the above.
2. Conventional therapy arm: Participants will receive standard treatment either at the hospital or from their general practitioner, without any influence from the trial and without starting trial-related medication.

Furthermore, a third group of 50 participants with coronary atherosclerosis and normal long-term average glucose levels will be included.

All trial participants will, at inclusion, be examined for the presence of diabetic nephropathy, diabetic neuropathy, diabetic retinopathy, and liver fat accumulation. This will be done through blood samples, urine samples, nerve examinations, and liver ultrasound. In addition, height, weight, waist circumference, body muscle and fat composition, pulse, and blood pressure will be measured. The third group will then conclude their participation.

The interventional therapy arm will begin the described intervention, which lasts for one year. After one year, the intervention period will end. Both randomized groups will then be examined by blood samples, urine samples, liver ultrasound, height, weight, waist circumference, body muscle and fat composition, pulse, and blood pressure. One year later, the above examinations will be repeated, except for the liver ultrasound. This will mark the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Chronic coronary syndrome with documented coronary artery disease. In the case of previous myocardial infarction, at least 30 days between the event and randomization is required.
* Prediabetes defined as HbA1c 42-47 mmol/mol (IEC criteria) OR normoglycemia defined as HbA1c <39 mmol/mol
* Age 18 to 80 years

Exclusion Criteria:

* eGFR <30 mL/min/1.73 m2
* Previous diabetes diagnosis, previous HbA1c >47 mmol/mol, or current/previous usage of diabetes medication
* Anemia, recent bleeding or blood transfusion (<3 months)
* Previous pancreatitis
* Pregnancy, breastfeeding, or fertile women who do not use highly effective contraception
* Strongly reduced liver function
* Chronic alcohol abuse
* Known hemoglobinopathy and other conditions with effect on erythrocyte lifespan
* Intake of medications with known effect on HbA1c validity such as: antiretroviral medications, trimethoprim, sulfamethoxazole, sulfasalazine hydroxyurea, dapsone, acetylsalicylic acid (>3 g/daily), high dose vitamin C and E.
* Heart failure with NYHA class III or IV Trial subjects must be capable of giving informed consent as assessed by the investigator.

Patients with BMI<25 kg/m2 will be assessed individually by an investigator for eligibility (e.g., whether initiation of a GLP-1 RA with potential weight loss is clinically justifiable).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Presence of a composite of retinopathy, nephropathy, neuropathy, and MASLD | Baseline
Incidence of normoglycemia defined as HbA1c <39 mmol/mol | 1-year follow-up

SECONDARY OUTCOMES:
Presence of: Retinopathy, Nephropathy, Neuropathy, or MASLD | Baseline
Presence of a composite of retinopathy, nephropathy, and neuropathy. | Baseline
Incidence of normoglycemia defined as HbA1c <42 mmol/mol | 1-year follow-up
Change in HbA1c | 1-year follow-up
Change in eGFR | 1-year follow-up
Change in cystatin-C | 1-year follow-up
Change in hs-CRP | 1-year follow-up
Change in lipid parameters | 1-year follow-up
Change in c-peptide | 1-year follow-up
Change in HOMA-IR | 1-year follow-up
Change in Fib-4 | 1-year follow-up
Change in CD163 | 1-year follow-up
Change in PRO-C3 | 1-year follow-up
Change in MASLD severity | 1-year follow-up
Change in urine albumin-creatinine ratio | 1-year follow-up
Change in weight | 1-year follow-up
Change in waist circumference | 1-year follow-up
Prevalence of HbA1c ≥42 mmol/mol | 2-year follow-up
  Main outcome of interest
Incidence of type 2 diabetes | 2-year follow-up
Prevalence of prediabetes defined as HbA1c 42-47 mmol/mol | 2-year follow-up
Prevalence of prediabetes defined as HbA1c 39-47 mmol/mol | 2-year follow-up
Change in HbA1c | 2-year follow-up
Change in eGFR | 2-year follow-up
Change in cystatin-C | 2-year follow-up
Change in hs-CRP | 2-year follow-up
Change in lipid parameters | 2-year follow-up
Change in c-peptide | 2-year follow-up
Change in HOMA-IR | 2-year follow-up
Change in Fib-4 | 2-year follow-up
Change in CD163 | 2-year follow-up
Change in PRO-C3 | 2-year follow-up
Change in weight | 2-year follow-up
Change in waist circumference | 2-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Michael Maeng, MD, PhD, Principal Investigator — Aarhus University Hospital, Department of Cardiology
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT07392151/Prot_SAP_000.pdf